CLINICAL TRIAL: NCT04786496
Title: Effects of Wise Interventions in Psychophysiological Responses to Stress
Brief Title: Wise Interventions and Responses to Stress
Acronym: ITP-RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Basque Country Government (Unknown); Spanish Government (Unknown)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ITP
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Stress, Physiological; Stress, Psychological; Social Stress; Depression
Keywords: Trier Social Stress Test; Social Stress; Stress reactivity; Heart Rate; Respiratory Sinus Arrhythmia; Skin Conductance Level; Cortisol; Mood; Young Adults
MeSH Terms: conditions — Stress, Psychological; Depression; Arrhythmia, Sinus

STUDY DESIGN:
Intervention Model Description: Participants were randomized (balanced for sex and levels of depression and social anxiety) to one of three groups (i.e., ITP+SA, ITP, and CC) in parallel for the duration of the study.
  Given the relevance of depression and social anxiety during stress tasks such as the TSST, these measures were used to balance participants within intervention and control groups. Specifically, a cluster analysis using mean scores on depression and social anxiety was conducted, resulting in a four-cluster solution according to the participants' level of depression and social anxiety. One-third of the males of each cluster and one-third of the females of each cluster were randomly assigned to each of the experimental conditions (i.e., ITP+SA, ITP, and CC). This allowed the three conditions to be balanced in gender and social anxiety and depression scores
Who Masked: Participant
Masking Description: Participants were blinded to the intervention condition. Moreover, both the speech and math tasks of the Trier Social Stress Test were done in front of two confederates (one woman and one man) who were blind to the intervention condition and who had not had previous contact with the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ITP+SA Wise intervention (Incremental Theory of Personality Intervention with Self-affirmations) (Experimental): Wise intervention (based on ITP and SA) consisting on several tasks to be completed individually. 30 minutes
  Interventions: Behavioral: ITP+SA Wise intervention
- ITP Wise intervention (Incremental Theory of Personality Intervention) (Experimental): Wise intervention (based on ITP) consisting on several tasks to be completed individually. 30 minutes
  Interventions: Behavioral: ITP Wise intervention
- Control Intervention (Other): Educational intervention (about heritage conservation) consisting on several tasks to be completed individually. 30 minutes
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: ITP+SA Wise intervention — Intervention designed to promote well-being and resilience in late adolescents and young adults. It includes two components: a self-affirmation (SA) activity and an ITP intervention. The SA component includes a list of values so that they could choose the three most important for them. Next, they are asked to write why those selected values are the most important to them. The ITP component resembled the intervention developed by David S. Yeager and colleagues and it was adapted to first year university students. It consisted of three parts. First, participants are asked to read scientific studies that provide evidence that behaviors are controlled pathways in the brain that have the potential to be changed under the right circumstances. Second, participants read several testimonials purportedly written by second year university students to bring credibility to the ITP. Finally, participants are asked to write their own version of such a narrative (self-persuasive writing exercise).
  Arms: ITP+SA Wise intervention (Incremental Theory of Personality Intervention with Self-affirmations)
Behavioral: ITP Wise intervention — Intervention designed to promote well-being and resilience in late adolescents and young adults based on four general types of change strategies: (1) scientific knowledge, (2) generation of new meanings, (3) commitment through action, and (4) active reflection. It includes the ITP component described above for the ITP+SA Wise intervention.
  Arms: ITP Wise intervention (Incremental Theory of Personality Intervention)
Behavioral: Control condition — The control intervention was designed to have a similar structure than the experimental interventions, including also reading and writing tasks, but that they were not in any way related to the contents of the experimental interventions. In particular, participants were asked to read an article about the fire that took place in the Notre Dame cathedral in Paris that had been recently published in a newspaper. Starting from the accident of the Notre Dame cathedral, the article focuses on reflecting on the problem of heritage conservation and analyzing the situation of other important cathedrals. After reading the article, the participants were asked to write a few lines evaluating in their opinion the importance of the conservation of historical buildings such as those mentioned and how much of the public economic budget should be used for heritage conservation.
  Arms: Control Intervention

SUMMARY:
This study compares the effects of two wise interventions (implicit theory of personality intervention and implicit theory of personality intervention plus self-affirmation) with a control condition in the stress responses of young adults. Responses include respiratory sinus arrhythmia, heart rate, skin conductance level, cortisol levels, and mood.

DETAILED DESCRIPTION:
Whereas several studies indicate that implicit theory of personality interventions (ITP) are promising in the prevention of depressive symptoms, evidence about the effects of the ITP intervention on stress pathways is scarce. The current study aims to elucidate the effects of ITP on psychophysiological responses to social stress in young adults during their transition to university. Based on preliminary findings that ITP was more effective among younger adolescents in reducing depressive symptoms and that a combination of ITP with self-affirmation (SA) was more effective in the prevention of other risky behaviors, the current study proposes that the addition of a SA component could increase the effectiveness of the ITP intervention when responding to stress. Thus, this study compares the effects of the ITP alone and in combination with a SA component in psychophysiological responses to a standardized social stressor (the Trier Social Stress Test, TSST). Both interventions (i.e., ITP+SA and ITP) are compared with a control condition (CC) in indicators of the autonomic nervous system (heart rate -HR-, respiratory sinus arrhythmia -RSA-, skin conductance level -SCL-), the hypothalamic-pituitary-adrenal axis (cortisol level), and subjective mood. The investigators expect that participants in both ITP interventions, and in ITP+SA intervention in particular, will display better stress responses during the stressful tasks compared with participants in the CC (i.e., lower HR and SCL increase, lower RSA suppression, and lower cortisol and negative mood increase). The investigators also expect that participants would display better recovery after the stressful tasks (i.e., higher HR and SCL decrease, and higher RSA increase).

Finally, this research will examine whether depressive symptoms moderate the effects of the intervention on stress responses. Previous research has shown that depression has been associated with dysregulated stress responses both at the autonomic nervous system and hypothalamic-pituitary-adrenal axis. Moreover, some studies have found that interventions are more effective among participants at risk to reduce both depression and stress. Therefore, the ITP intervention, alone and in combination with SA, could be more beneficial among those participants with higher levels of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the participants.
* To be fluent in Spanish.

Exclusion criteria:

* Having cardiovascular disease.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline levels of cortisol in saliva at recovery (immediately after the procedure -Trier Social Stress Task-). | Baseline and immediately after the math phase of the Trier Social Stress Task.
  Participants provided saliva samples to be assayed for neuroendocrine levels to measure cortisol. They were directed to transfer saliva from their mouths to a tube. The sample tubes were carefully labelled and stored in a freezer at -25 ºC until they were sent to the Medikosta Laboratory.
Change from baseline levels of heart-rate (HR) at the time of the procedure (i.e., during the Trier Social Stress Task) and recovery (i.e., immediately after the Trier Social Stress Task). | Baseline, during the procedure, and immediately after the procedure (i.e., the Trier Social Stress Task).
  Electrocardiogram (ECG) to measure heart-rate (HR) was recorded using the BioPac M150 system at a sampling rate of 1000 Hz and AcqKnowledge® 4.0 software.
Change from baseline levels of heart-rate variability (HRV) at the time of the procedure (i.e., during the Trier Social Stress Task) and recovery (i.e., immediately after the Trier Social Stress Task). | Baseline, during the procedure, and immediately after the procedure (i.e., the Trier Social Stress Task).
  Electrocardiogram (ECG) to measure heart-rate variability (HRV) was recorded using the BioPac M150 system at a sampling rate of 1000 Hz and AcqKnowledge® 4.0 software.
Change from baseline levels of skin conductance level (SCL) at the time of the procedure (i.e., during the Trier Social Stress Task) and recovery (i.e., immediately after the Trier Social Stress Task). | Baseline, during the procedure, and immediately after the procedure (i.e., the Trier Social Stress Task).
  Electrodermal Activity to measure skin conductance level (SCL) was recorded using the BioPac M150 system at a sampling rate of 1000 Hz and AcqKnowledge® 4.0 software.
Change from baseline scores of the subscale for Negative Mood of the Scale for Mood Assessment (Sanz, 2001) at recovery (immediately after the procedure -Trier Social Stress Task-). | Baseline and immediately after the math phase of the Trier Social Stress Task.
  Self reported transitory negative moods measured by 12 items (assessing depression, anxiety, and hostility) scored on an 11-point scale from 0 (nothing) to 10 (a lot), yielding a total between 0 and 120 (with higher scores meaning higher negative moods).
Change from baseline scores of the subscale for Positive Mood of the Scale for Mood Assessment (Sanz, 2001) at recovery (immediately after the procedure -Trier Social Stress Task-). | Baseline and immediately after the math phase of the Trier Social Stress Task.
  Self reported transitory positive mood measured by 4 items (assessing elation) scored on an 11-point scale from 0 (nothing) to 10 (a lot), yielding a total between 0 and 40 (with higher scores meaning higher positive mood).

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at OSF when the results of the study are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent protocol will be published at clinicaltrials.org Data will be available at OSF when the results are published.
Access Criteria: Public